CLINICAL TRIAL: NCT06637696
Title: The Effect of Implementation of Bundle for Preventing Blood Culture Contamination in Neonatal Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Oğuz Han Kalkanlı, Medical Doctor, Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: BU-OK-01
Record Dates: First submitted 2024-10-01; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Newborn; Infection
Keywords: blood culture bundle; blood culture contamination; cost-effectiveness; neonatal intensive care unit; neonates
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: The study included a total of 320 (160 neonates in pre-bundle period, 160 neonates in post-bundle period) neonates.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Culture Bundle Group (Active Comparator): In this group, blood culture collection was performed using a checklist other than the standard criteria.The checklist for the blood culture contamination precaution package (Table 1) was prepared using guidelines from the Turkish Society of Clinical Microbiology.
  Interventions: Other: Blood Culture Bundle
- Control Blood Culture Group (Placebo Comparator): In this group the standard practice in both periods was aseptic, non-contact technique for blood culture collection. For this purpose, hands were cleaned with antibacterial liquid soap (Klorhexin scrub antibacterial liquid soap 4-% Ekin Medical), the patient's skin was cleaned with povidone iodine 10% solution (Betadix 10% solution- Natural Medical Pharma) using sterile gloves, waited at least 30 seconds and then povidone iodine was removed from the skin with 70% alcohol.
  Interventions: Other: Blood Culture Bundle

INTERVENTIONS:
Other: Blood Culture Bundle — In this pre and post intervention study investigators aimed to evaluate the impact of a blood culture bundles on the incidence of blood culture contamination rates in NICU.

SUMMARY:
In this study, investigators aimed to evaluate the impact of blood culture bundles on the incidence of contamination in the neonatal intensive care unit (NICU).

DETAILED DESCRIPTION:
Infections are never as frequent and life-threatening as in the neonatal period. The lack of sepsis-specific findings in the neonatal period, the narrow repertoire of clinical findings in newborns, and the fact that non-infectious clinical conditions frequently encountered in this period have similar findings pose a serious problem for early diagnosis and treatment of neonatal sepsis. Another important problem is that early empirical antibiotic treatment without diagnostic confirmation has to be resorted to very frequently in order to avoid morbidity and more importantly mortality with early intervention. This leads to unnecessary and prolonged treatment of newborns with potentially dangerous broad-spectrum antibiotics as well as prolonged hospitalizations and significant costs.

The rate of contaminated blood culture in the neonatal period is 2.6-18%. In this study, investigators aimed to evaluate the impact of blood culture bundles on the incidence of contamination in the neonatal intensive care unit (NICU).

ELIGIBILITY:
Inclusion Criteria:

Newborns diagnosed with sepsis

Exclusion Criteria:

Newborns receiving antibiotic treatment

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Blood Culture Contamination Rate | 1 year
  The primary purpose of this study is to compare the contamination rate of blood culture taken with the bundle method and the contamination rate of blood culture taken with the standard method.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Han Kalkanlı, Principal Investigator — Dr. Behcet Uz Children's Hospital
Locations (1):
- Dr. Behcet Uz Children's Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No